CLINICAL TRIAL: NCT01485289
Title: Stabilimax Study Participants Collection of Additional Follow-up Data Clinical Investigation Plan R-001
Brief Title: Stabilimax Investigational Device Exemption (IDE) Clinical Investigation Patient Followup Study
Status: Completed | Type: Observational
Sponsor: Rachiotek LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MLucey
Record Dates: First submitted 2011-09-29; First posted 2011-12-05 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Investigational Stabilimax
- Control, Posterolateral Fusion

SUMMARY:
The intent of this study is to complete the collection of clinical data on subjects enrolled in the Stabilimax Dynamic Spine Stabilization IDE clinical trial (#G060214) sponsored by the now defunct Applied Spine Technologies Inc . The Applied Spine assets, including the clinical trial data, were acquired by Rachiotek, LLC in 2010. When Applied Spine ceased their funding of the trial, a number of enrolled patients had not yet completed the two year follow-up visit defined as the study endpoint in the clinical investigation plan. No additional patient treatment is required to complete the study. Rachiotek has interest in pursuing IDE approval for a new study and the information collected in this study is essential for supporting the new Investigational Device Exemption application.

ELIGIBILITY:
Inclusion Criteria:

* Any patient that after having met all of the inclusion/exclusion criteria identified for the Stabilimax Investigational Device Exemption study had enrolled in the Stabilimax Investigational Device Exemption study and were implanted with the Stabilimax NZ or the control device.

Exclusion Criteria:

* Any patient that has had the device removed and the adverse event follow-up report stated that the event was resolved. This applies only if the patient was formally withdrawn from the study at that time.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2011-08; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) for Leg Pain | Minimum 24 months post procedure
  Patient demonstrates a reduction in leg pain from baseline of at least 20 mm on a 100 mm visual analog scale (VAS)
Zurich Claudication Questionnaire (ZCQ) | Minimum 24 months post procedure
  Clinically significant improvement from baseline defined by a minimum decrease of .5 as measured by the Zurich Claudication Questionnaire for both Symptom Severity(SS) and Physical Function (PF) scores
Major Device Related (MDR) Complications | Minimum 24 months post procedure
  Patient experiences no major device-related complications
Revision, Reoperation, or Removal | Minimum 24 months post procedure
  The treated level did not require surgical revision, reoperation, removal, or supplemental fixation.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | Minimum 24 months post procedure
  Changes from baseline in function scores (Oswestry Disability Index)
Presence (control) or Absence (Stabilimax)of fusion | Minimum 24 months post procedure
  Presence (control patients) or absence (Stabilimax NZ® patients) of fusion at 24-months post procedure
Adverse Events (AE) | Minimum 24 months post procedure
  safety will be assessed by quantification of the incidence of all adverse events observed during the study period by type.
Physician Satisfaction Scale | Immediately post procedure
  Characterization of the physician's satisfaction with clinical implantation of the therapeutic device by use of rating scales.

CONTACTS AND LOCATIONS:
Locations (1):
- Triangle Orthopedics, Durham, North Carolina, United States